CLINICAL TRIAL: NCT03232281
Title: A Phase III, Multicentre, Randomised, Open-label, Parallel, Active-controlled Study to Compare the Oestradiol Suppression, Clinical Efficacy and Safety of Two Formulations of Triptorelin (Triptorelin Pamoate PR 3-month and Triptorelin Acetate PR 1-month) in Chinese Subjects With Endometriosis
Brief Title: Study to Compare the Oestradiol Suppression, Clinical Efficacy and Safety of Two Formulations of Triptorelin (Triptorelin Pamoate PR 3-month and Triptorelin Acetate PR 1-month) in Chinese Subjects With Endometriosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-CN-52014-220
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Triptorelin Pamoate; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triptorelin pamoate PR 3-month (Experimental): Subjects received 15 mg triptorelin pamoate per injection, administered as an intramuscular injection once every 12 weeks (a total of 2 injections, at baseline and Week 12).
  Interventions: Drug: Triptorelin Pamoate PR 3-month
- Triptorelin acetate PR 1-month (Active Comparator): Subjects received 3.75 mg triptorelin acetate per injection, administered as an intramuscular injection once every 4 weeks (a total of 6 injections, at baseline and Weeks 4, 8, 12, 16 and 20).
  Interventions: Drug: Triptorelin Acetate PR 1-month

INTERVENTIONS:
Drug: Triptorelin Pamoate PR 3-month — 15mg/injection, administered as an intramuscular injection once every 12 weeks (a total of 2 injections).
  Other Names: Triptorelin pamoate for injection 15 mg
  Arms: Triptorelin pamoate PR 3-month
Drug: Triptorelin Acetate PR 1-month — 3.75mg/injection, administered as an intramuscular injection once every 4 weeks (a total of 6 injections)
  Other Names: Diphereline 3.75 mg
  Arms: Triptorelin acetate PR 1-month

SUMMARY:
To assess the efficacy of triptorelin pamoate prolonged release (PR) 3-month formulation in Chinese female subjects with endometriosis by demonstrating the non-inferiority of triptorelin pamoate PR 3-month formulation injected once as compared to triptorelin acetate PR 1-month formulation injected 3 times consecutively.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged from 18 to 45 years inclusive at the date of informed consent.
* A history of active and regular menstrual cycles of 21 to 35 days (inclusive) in the 6 months prior to the screening visit.
* A diagnosis of endometriosis, confirmed by laparoscopy or laparotomy within10 years prior to the screening visit.
* Requires treatment with a Gonadotrophin releasing hormone (GnRH) agonist for a period of 6 months in the judgement of the investigator.

Exclusion Criteria:

* A current history of undiagnosed abnormal genital bleeding.
* Received treatment with a GnRH agonist within 6 months prior to the screening visit.
* Received any other hormonal treatment within 3 months prior to the screening visit (oestrogens, progestogens, danazol, gestrinone and cyproterone acetate etc).
* Chronic pelvic pain that is not caused by endometriosis, that would interfere with the assessment of endometriosis-associated pelvic pain.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (24):
- China (24):
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Hainan General Hospital, Haikou
  - Women's Hospital, School of Medicine Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital school of medicine, Zhejiang University, Hangzhou
  - Nanjing Maternity and Child Health Care Hospital, Nanjing
  - Zhongda Hospital, Southeast University, Nanjing
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Obstetrics and Gynaecology Hospital of Fudan University, Shanghai
  - Shanghai Tongji Hospital, Shanghai
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Medical University General Hospital, Tianjin
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Northern Jiangsu People's Hospital, Yangzhou
  - General Hospital of Ningxia Medical University, Yinchuan

REFERENCES:
- [Derived] Li X, Li H, Shi H, Li X, Zhou R, Lu D, Cai Y, Zhou Y, Cabri P, Shi X, Pedret-Dunn A, Leng J. Assessment of Two Formulations of Triptorelin in Chinese Patients with Endometriosis: A Phase 3, Randomized Controlled Trial. Adv Ther. 2022 Oct;39(10):4663-4677. doi: 10.1007/s12325-022-02264-5. Epub 2022 Aug 10. PMID 35947347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female subjects aged from 18 to 45 years were recruited to this Phase 3 randomised, open-label study at 24 study centres in China between 28 July 2017 and 16 November 2019.
Pre-assignment Details: Subjects who met the inclusion criteria and none of the exclusion criteria were randomised in a 1:1 ratio, stratified according to endometriotic surgical history and the severity of endometriosis-associated pelvic pain.
Groups:
- Triptorelin Pamoate PR 3-month: Subjects received 15 milligrams (mg) triptorelin pamoate per injection, administered as an intramuscular (IM) injection once every 12 weeks (a total of 2 injections, at baseline and Week 12).
- Triptorelin Acetate PR 1-month: Subjects received 3.75 mg triptorelin acetate per injection, administered as an IM injection once every 4 weeks (a total of 6 injections, at baseline and Weeks 4, 8, 12, 16 and 20).
Period: Overall Study
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month
Started | 150 | 150
Received Treatment | 149 | 150
Completed Week 12 | 143 | 148
Completed Week 24 | 143 | 144
Completed | 143 | 144
Not Completed | 7 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Protocol Deviation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the randomised set.
Groups:
- Triptorelin Pamoate PR 3-month: Subjects received 15 mg triptorelin pamoate per injection, administered as an IM injection once every 12 weeks (a total of 2 injections, at baseline and Week 12).
- Total: Total of all reporting groups
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (6.1) | 32.6 (6.2) | 32.5 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 150 | 300
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 150 | 150 | 300
  Not Hispanic or Latino | 150 | 150 | 300
Region of Enrollment [Number; unit: participants]
  China | 150 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Castrated (E2 ≤184 Pmol/L or 50 pg/mL) at Week 12
Description: Castration was defined as serum oestradiol (E2) ≤184 picomoles/litre (pmol/L) or 50 picograms/millilitre (pg/mL).
  The primary endpoint was evaluated based on centralised blinded bioanalysis of serum samples for E2. The percentage of subjects castrated and the 95% asymptotic confidence intervals (CIs), calculated from binomial distribution, are presented.
Time Frame: Week 12
Population: The per protocol set included all randomised subjects who received at least one dose of study medication with at least one baseline and at least one post-baseline assessment of the primary efficacy parameter, and without major protocol violations/deviations affecting the primary efficacy endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month
Number analyzed (Participants) | 142 | 146
percentage of subjects | 98.6 [96.65 to 100.00] | 99.3 [97.98 to 100.00]
Statistical Analysis 1: Comparison: Triptorelin Pamoate PR 3-month vs Triptorelin Acetate PR 1-month; The null hypothesis was that triptorelin pamoate PR 3-month was inferior to triptorelin acetate PR 1-month. The alternative hypothesis was that triptorelin pamoate PR 3-month was non-inferior to triptorelin acetate PR 1-month; Test type: Non-Inferiority — If the lower limit of the 95% CI for the difference was >-10%, triptorelin pamoate PR 3-month non-inferiority to triptorelin acetate PR 1-month was confirmed; Rate difference (%) = -0.7, 95% CI 2-sided [-4.41 to 2.58] — The rate difference (triptorelin pamoate PR 3-month - triptorelin acetate PR 1-month) and the 2-sided 95% CI of the difference were calculated using the Miettinen and Nurminen method, stratified by randomisation stratification factors

2. Secondary Outcome: Percentage of Subjects Castrated (E2 ≤184 Pmol/L or 50 pg/mL) at Weeks 4 and 8
Description: The percentages of subjects who were castrated at Weeks 4 and 8 where castration was defined as serum E2 ≤184 pmol/L or 50 pg/mL are presented. The 95% asymptotic CIs were calculated from the binomial distribution.
Time Frame: Weeks 4 and 8
Population: The full analysis set included all randomised subjects who received at least one dose of study medication with at least one baseline and at least one post-baseline assessment of the primary efficacy parameter.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month
Number analyzed (Participants) | 147 | 150
percentage of subjects
  Week 4 | 98.0 [95.67 to 100.00] | 99.3 [98.03 to 100.00]
  Week 8 | 97.3 [94.65 to 99.91] | 100.0 [100.00 to 100.00]
Statistical Analysis 1: Comparison: Triptorelin Pamoate PR 3-month vs Triptorelin Acetate PR 1-month; Rate difference at Week 4. The null hypothesis was that triptorelin pamoate PR 3-month was inferior to triptorelin acetate PR 1-month. The alternative hypothesis was that triptorelin pamoate PR 3-month was non-inferior to triptorelin acetate PR 1-month; Test type: Non-Inferiority — If the lower limit of the 95% CI for the difference was >-10%, triptorelin pamoate PR 3-month non-inferiority to triptorelin acetate PR 1-month was observed without multiplicity adjustment; Rate difference (%) = -1.3, 95% CI 2-sided [-5.26 to 1.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Triptorelin Pamoate PR 3-month vs Triptorelin Acetate PR 1-month; Rate difference at Week 8. The null hypothesis was that triptorelin pamoate PR 3-month was inferior to triptorelin acetate PR 1-month. The alternative hypothesis was that triptorelin pamoate PR 3-month was non-inferior to triptorelin acetate PR 1-month; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Rate difference (%) = -2.7, 95% CI 2-sided [-6.80 to -0.16] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Subjects Castrated (E2 ≤110 Pmol/L or 30 pg/mL) at Weeks 4, 8 and 12
Description: The percentages of subjects who were castrated at Weeks 4, 8 and 12 where castration was defined as serum E2 ≤110 pmol/L or 30 pg/mL are presented. The 95% asymptotic CIs were calculated from the binomial distribution.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month
Number analyzed (Participants) | 147 | 150
percentage of subjects
  Week 4 | 98.0 [95.67 to 100.00] | 99.3 [98.03 to 100.00]
  Week 8 | 95.2 [91.80 to 98.68] | 99.3 [98.03 to 100.00]
  Week 12 | 95.9 [92.72 to 99.12] | 98.7 [96.83 to 100.00]
Statistical Analysis 1: Comparison: Triptorelin Pamoate PR 3-month vs Triptorelin Acetate PR 1-month; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Rate difference (%) = -1.3, 95% CI 2-sided [-5.26 to 1.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Triptorelin Pamoate PR 3-month vs Triptorelin Acetate PR 1-month; [analysis description as in outcome 2, analysis 2]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Rate difference (%) = -4.1, 95% CI 2-sided [-8.93 to -0.52] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Triptorelin Pamoate PR 3-month vs Triptorelin Acetate PR 1-month; Rate difference at Week 12. The null hypothesis was that triptorelin pamoate PR 3-month was inferior to triptorelin acetate PR 1-month. The alternative hypothesis was that triptorelin pamoate PR 3-month was non-inferior to triptorelin acetate PR 1-month; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Rate difference (%) = -2.7, 95% CI 2-sided [-7.44 to 1.17] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Endometriosis-associated Pelvic Pain at Weeks 4, 8 and 12
Description: Endometriosis-associated pelvic pain was assessed using a 100 millimetres (mm) visual analogue scale (VAS) where subjects indicated the subjective level of their most severe endometriosis pain over the last 4 weeks by making a single vertical mark on the line ranging from 'absence of pain' (0 mm) to 'unbearable pain' (100 mm). Lower scores indicated a better outcome. Baseline was defined as the last available assessment prior to the first dose of study medication. The least squares (LS) mean change from baseline at each timepoint as measured by the VAS is presented.
Time Frame: Baseline (Day 1) and Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month
Number analyzed (Participants) | 147 | 150
mm
  Week 4: number analyzed (Participants) | 147 | 149
  Week 4 | -24.4 [-27.2 to -21.6] | -24.4 [-27.1 to -21.6]
  Week 8: number analyzed (Participants) | 146 | 150
  Week 8 | -28.5 [-31.1 to -25.9] | -27.8 [-30.3 to -25.2]
  Week 12: number analyzed (Participants) | 146 | 148
  Week 12 | -28.1 [-30.6 to -25.7] | -28.4 [-30.8 to -26.0]

5. Secondary Outcome: Mean E2 Concentration at Weeks Baseline and 4, 8 and 12
Description: The mean serum E2 concentrations at baseline and Weeks 4, 8 and 12 are presented.
Time Frame: Baseline (Day 1) and Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month
Number analyzed (Participants) | 147 | 150
pmol/L
  Baseline | 192.302 (258.209) | 218.893 (296.825)
  Week 4 | 25.347 (46.253) | 18.959 (3.944)
  Week 8: number analyzed (Participants) | 146 | 150
  Week 8 | 47.175 (156.521) | 21.863 (12.550)
  Week 12: number analyzed (Participants) | 146 | 148
  Week 12 | 36.600 (76.882) | 26.695 (31.174)

6. Secondary Outcome: Mean Follicle Stimulating Hormone (FSH) Concentration at Baseline and Weeks 4, 8 and 12
Description: The mean FSH concentrations at baseline and Weeks 4, 8 and 12 are presented.
Time Frame: Baseline (Day 1) and Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International Units/L (IU/L)
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month
Number analyzed (Participants) | 147 | 150
International Units/L (IU/L)
  Baseline | 6.099 (3.929) | 6.258 (4.520)
  Week 4: number analyzed (Participants) | 147 | 149
  Week 4 | 1.762 (1.373) | 1.699 (1.049)
  Week 8: number analyzed (Participants) | 146 | 150
  Week 8 | 2.891 (1.163) | 2.766 (1.329)
  Week 12: number analyzed (Participants) | 146 | 148
  Week 12 | 3.344 (1.347) | 3.325 (1.414)

7. Secondary Outcome: Mean Luteinising Hormone (LH) Concentration at Baseline and Weeks 4, 8 and 12
Description: The mean LH concentrations at baseline and Weeks 4, 8 and 12 are presented.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month
Number analyzed (Participants) | 147 | 150
IU/L
  Baseline | 3.376 (1.902) | 3.487 (1.858)
  Week 4: number analyzed (Participants) | 147 | 149
  Week 4 | 0.660 (1.771) | 0.500 (0.173)
  Week 8: number analyzed (Participants) | 146 | 150
  Week 8 | 0.444 (1.928) | 0.255 (0.122)
  Week 12: number analyzed (Participants) | 146 | 148
  Week 12 | 0.324 (0.555) | 0.251 (0.239)

8. Secondary Outcome: Median Time to Menses Recovery
Description: Time to menses recovery was defined as the time (in days) between the date of the last dose of study medication and the date of the first day the subject observed menstrual bleeding of the next menstrual period. Menses recovery status was assessed at all study visits from Day 1 to the end of study visit. The median time to menses recovery was analysed using the Kaplan-Meier method.
Time Frame: Baseline (Day 1) up to Week 40 (end of study visit)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month
Number analyzed (Participants) | 147 | 150
days | 179.0 [172.0 to 182.0] | 85.0 [82.0 to 87.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were monitored from Day 1 up to Week 28 (approximately 7 months).
Description: A TEAE was defined as any adverse event that occurred or worsened on or after the first dose, through 112 days (16 weeks) after last injection of triptorelin pamoate PR 3-month or through 56 days (8 weeks) after last injection for triptorelin acetate PR 1-month. TEAEs are presented for the safety set which included all subjects who received at least one dose of study medication.
Arm/Group | Triptorelin Pamoate PR 3-month | Triptorelin Acetate PR 1-month
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/150
Serious Adverse Events (participants affected / at risk) | 2/149 | 1/150
Other Adverse Events (participants affected / at risk) | 132/149 | 135/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate PR 3-month (N=149) | Triptorelin Acetate PR 1-month (N=150)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate PR 3-month (N=149) | Triptorelin Acetate PR 1-month (N=150)
Abdominal pain lower (Gastrointestinal disorders) | 4 (4) | 13 (19)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 4 (4)
Pyrexia (General disorders) | 6 (6) | 8 (9)
Nasopharyngitis (Infections and infestations) | 16 (19) | 24 (30)
Upper respiratory tract infection (Infections and infestations) | 37 (46) | 27 (34)
Vaginal infection (Infections and infestations) | 8 (9) | 7 (7)
Protein urine present (Investigations) | 9 (9) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (19) | 13 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 9 (13)
Dizziness (Nervous system disorders) | 6 (7) | 9 (11)
Headache (Nervous system disorders) | 10 (11) | 9 (11)
Insomnia (Psychiatric disorders) | 14 (14) | 8 (8)
Menorrhagia (Reproductive system and breast disorders) | 11 (13) | 6 (6)
Vaginal haemorrhage (Reproductive system and breast disorders) | 66 (79) | 68 (82)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (9)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 (10) | 12 (12)
Night sweats (Skin and subcutaneous tissue disorders) | 19 (20) | 13 (13)
Hot flush (Vascular disorders) | 86 (90) | 89 (91)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT03232281/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT03232281/SAP_001.pdf